CLINICAL TRIAL: NCT05862779
Title: Effects of Omega-3 and Whey Protein Supplementation on Lean Mass and Strength Gains in Older Adults Performing Resistance Exercise: A Randomized, Double-Blind and Placebo-Controlled Study
Brief Title: Effects of Omega-3 and Whey Protein Supplementation on Lean Mass in Older Adults
Acronym: W-3 and Whey
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Erick Prado de Oliveira, Assistant professor, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5.728.049
Record Dates: First submitted 2023-04-10; First posted 2023-05-17 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Whey Proteins; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Group (Placebo Comparator): Group supplemented with maltodextrin (40g/day) and corn oil (4g/day). All groups will undergo a training program with strength exercises for 12 weeks
  Interventions: Dietary Supplement: Placebo Group
- Whey Protein + Placebo (Experimental): Group supplemented with isolated whey protein (40g/day) and corn oil (4g/day). All groups will undergo a training program with strength exercises for 12 weeks.
  Interventions: Dietary Supplement: Whey Protein + Placebo
- Omega 3 + Placebo (Experimental): Group supplemented with omega-3 (4g/day) and maltodextrin (40g/day). All groups will undergo a training program with strength exercises for 12 weeks.
  Interventions: Dietary Supplement: Omega 3 + Placebo
- Omega 3 + Whey Protein (Experimental): Group supplemented with omega-3 (4g/day) and whey protein (40g/day). All groups will undergo a training program with strength exercises for 12 weeks.
  Interventions: Dietary Supplement: Omega 3 + Whey Protein

INTERVENTIONS:
Dietary Supplement: Placebo Group — The placebo group will receive 4 g per day of corn oil and 40 g per day of maltodextrin.
  Arms: Placebo Group
Dietary Supplement: Whey Protein + Placebo — The whey protein + placebo group will receive 40g per day of whey and 4g per day of corn oil.
  Arms: Whey Protein + Placebo
Dietary Supplement: Omega 3 + Placebo — The omega 3 + placebo group will receive 4 g per day of fish oil and 40 g per day of maltodextrin.
  Arms: Omega 3 + Placebo
Dietary Supplement: Omega 3 + Whey Protein — The omega 3 + whey group will receive 4g per day of fish oil and 40g per day of protein.
  Arms: Omega 3 + Whey Protein

SUMMARY:
To evaluate the effect of omega-3 supplementation combined with whey protein intake on lean mass and strength gains in older adults performing resistance exercise. Participants will be randomized into the 4 groups. The placebo group will receive 4 g per day of corn oil and 40 g per day of maltodextrin. The omega 3 + placebo group will receive 4 g per day of fish oil and 40 g per day of maltodextrin. The whey protein + placebo group will receive 40g per day of whey and 4g per day of corn oil. The omega 3 + whey group will receive 4g per day of fish oil and 40g per day of protein. All will perform the same exercise protocol for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (at least 1 year of menstrual interruption, self-reported);
* To be able to practice strength exercises;
* To be able to carry out supplementation;
* Do not present physical, orthopedic or cardiovascular complications that prevent the performance of physical exercises;
* No history of stroke or acute myocardial infarction;
* Not being a smoker and/or alcoholic;
* Do not perform hormone replacement therapy;
* Do not use anti-inflammatory drugs;
* To have normal kidney function;
* To submit a medical certificate of health that proves that the individual is able to perform exercises.

Exclusion Criteria:

* Do not provide the necessary information for the development of the study;
* Individuals with diseases previously diagnosed and undergoing treatment, such as type II diabetes mellitus, cancer, rheumatoid arthritis, high blood pressure, dyslipidemia, cardiovascular, and kidney and/or liver diseases.

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Changes in lean mass (kg) using ultrasound and electrical bioimpedance in postmenopausal women | up to 12 weeks

SECONDARY OUTCOMES:
Changes in strength (kg) using dynamometer in postmenopausal women | up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No